CLINICAL TRIAL: NCT04803760
Title: Evaluation of the Relationship Between Neck Pain and Ergonomic Factors in Office Workers
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Istanbul Physical Medicine and Rehabiltation Training and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Cansin Medin Ceylan, specialist, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: 2021/18
Record Dates: First submitted 2021-03-14; First posted 2021-03-18 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Disability Physical; Neck Pain; Ergonomic Factors
Keywords: neck pain; office workers; ergonomic factors
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mild disability: Those whose neck disability index value is 25 and below
  Interventions: Other: A self-administered questionnaire
- high disability: Those whose neck disability index value is 25 and above
  Interventions: Other: A self-administered questionnaire

INTERVENTIONS:
Other: A self-administered questionnaire — A self-administered questionnaire will be used to screen Neck disability index, demographic information and ergonomic risk factors.

SUMMARY:
Neck pain is a prevalent condition and leading causes of disability particularly in office workers compared to other occupations (1-3). Neck pain is not only a risk factor for functional disability but it is also associated with decreased productivity of workers and quality of life (4). However, the present literature is insufficient to determine the factors affecting the level of disability caused by neck pain among office workers where intensive computer use is common (5). Thus, the current study aimed to explore the associations between disability levels and of occupational risk factors in computer-using office workers with neck pain.

DETAILED DESCRIPTION:
This is a cross-sectional study. All participants will provide informed consent before participating in the study. The study will be conducted in accordance with the Helsinki Declaration criteria. Data will be collected using questionnaires, which include the Neck disability index, demographic information (including age, gender, educational level) and frequency of neck and head pain, history of general neck injuries and treatments applied. Also, years of office work at current job, sick leave, ergonomic training, duration of computer use per day and using of headphones, monitor and keyboard stand, mouse/mouse pad and number of computer screens will be determined.

In addition, based on Rapid Office Strain Assessment (ROSA) method the potential ergonomic risk factors computer position, computer screen position, head and back position and mouse position will be determined. Visual pictures of the work positions will be shown to the participants and the participants will be asked to select the appropriate pictures showing their work positions.

A self-administered questionnaire will be used to screen potential participants for this study. Inclusion criteria are individuals aged between 18 and 55, working on computer, having neck pain at least three months.

Exclusion criteria are reporting pregnancy, having a history of accidents, trauma or surgery in the neck region, congenital anomaly of the spine, rheumatologic disease, osteoporosis, spondylosis, spondylolisthesis, infection of the spine and discs, tumor.

Patients will be divided into 3 groups as mild, moderate and severe disabled according to their neck disability index values and will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 55,
* working on computer,
* having neck pain at least three months.

Exclusion Criteria:

* reporting pregnancy,
* having a history of accidents,
* trauma or surgery in the neck region,
* congenital anomaly of the spine,
* rheumatologic disease,
* osteoporosis,
* spondylosis,
* spondylolisthesis,
* infection of the spine
* cervical disc herniation,
* tumor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: aged between 18 and 55, working on computer, having neck pain at least three months.
Sampling Method: Non-Probability Sample
Enrollment: 1028 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
neck disability index | baseline
  The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain

CONTACTS AND LOCATIONS:
Overall Officials: cansın medin-ceylan, M.D., Principal Investigator — istanbul physical medicine rehabilitation research and training hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cote P, van der Velde G, Cassidy JD, Carroll LJ, Hogg-Johnson S, Holm LW, Carragee EJ, Haldeman S, Nordin M, Hurwitz EL, Guzman J, Peloso PM; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. The burden and determinants of neck pain in workers: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S60-74. doi: 10.1097/BRS.0b013e3181643ee4. PMID 18204402
- [Background] Aas RW, Tuntland H, Holte KA, Roe C, Lund T, Marklund S, Moller A. Workplace interventions for neck pain in workers. Cochrane Database Syst Rev. 2011 Apr 13;2011(4):CD008160. doi: 10.1002/14651858.CD008160.pub2. PMID 21491405
- [Background] Vassilaki M, Hurwitz EL. Insights in public health: perspectives on pain in the low back and neck: global burden, epidemiology, and management. Hawaii J Med Public Health. 2014 Apr;73(4):122-6. No abstract available. PMID 24765562
- [Background] Matsudaira K, Kawaguchi M, Isomura T, Inuzuka K, Koga T, Miyoshi K, Konishi H. Assessment of psychosocial risk factors for the development of non-specific chronic disabling low back pain in Japanese workers-findings from the Japan Epidemiological Research of Occupation-related Back Pain (JOB) study. Ind Health. 2015;53(4):368-77. doi: 10.2486/indhealth.2014-0260. Epub 2015 Jun 6. PMID 26051289
- [Background] McLean SM, May S, Klaber-Moffett J, Sharp DM, Gardiner E. Risk factors for the onset of non-specific neck pain: a systematic review. J Epidemiol Community Health. 2010 Jul;64(7):565-72. doi: 10.1136/jech.2009.090720. Epub 2010 May 12. PMID 20466711